CLINICAL TRIAL: NCT00660894
Title: Randomized Phase III Study of UFT+Leucovorin vs. TS-1 as Adjuvant Treatment for Stage III Colon Cancer , and Investigate Predictive Factors Based on Gene Expression
Brief Title: Tegafur-Uracil and Leucovorin or S-1 in Treating Patients With Stage III Colon Cancer That Has Been Completely Removed by Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000593164; TMDU-TRICC0706 (Other: National Cancer Institute)
Record Dates: First submitted 2008-04-16; First posted 2008-04-17 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Colorectal Cancer
Keywords: adenocarcinoma of the colon; stage III colon cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Leucovorin; Tegafur; S 1 (combination); titanium silicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- tegafur-gimeracil-oteracil potassium (Experimental): Patients receive tegafur-gimeracil-oteracil potassium(S-1) orally twice daily for 28 days with a subsequent pause of 14 days. This repeats 4 times every 6 weeks.
  Interventions: Drug: tegafur-gimeracil-oteracil potassium
- tegafur-uracil and folinate calcium (Active Comparator): Patients receive tegafur-uracil(UFT) plus folinate calcium(leucovorin) orally every 8 hours for 21 days with a subsequent pause of 7 days. This repeats 5 times every 5 weeks.
  Interventions: Drug: folinate calcium; Drug: tegafur-uracil

INTERVENTIONS:
Drug: folinate calcium
  Other Names: Leucovorin, leucovorin
  Arms: tegafur-uracil and folinate calcium
Drug: tegafur-uracil
  Other Names: UFT
  Arms: tegafur-uracil and folinate calcium
Drug: tegafur-gimeracil-oteracil potassium
  Other Names: S-1, TS-1
  Arms: tegafur-gimeracil-oteracil potassium

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as tegafur-uracil, leucovorin, and S-1, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. It is not yet known whether giving tegafur-uracil together with leucovorin is more effective than giving S-1 in treating patients with stage III colon cancer.

PURPOSE: This randomized phase III trial is studying giving tegafur-uracil together with leucovorin to see how well it works compared with giving S-1 in treating patients with stage III colon cancer that has been completely removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the disease-free survival of patients with stage III colon cancer treated with S-1 or tegafur-uracil and leucovorin after curative surgery .

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral tegafur-uracil and oral leucovorin 3 times daily on days 1-21. The treatment repeats 5 times every 5 weeks.
* Arm II: Patients receive oral S-1 twice daily on days 1-28. The treatment repeats 4 times every 6 weeks.

Biological samples are collected for gene expression analysis for identification of predictive markers.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of colon

  * Stage III (T1-4, N1-3, M0) disease
* Has undergone surgical resection of the tumor within the past 8 weeks

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Able to take medications orally
* WBC ≥ 3,500/mm³ and < 12,000/mm³
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9.0 g/dL
* Total bilirubin ≤ 2.0 mg/dL
* AST/ALT ≤ 100 IU/L
* Creatinine ≤ 1.2 mg/dL
* No other active malignancies
* Must have none of the following comorbidities:

  * Severe postoperative complications
  * Uncontrollable diabetes mellitus
  * Uncontrollable hypertension
  * Myocardial infraction within 6 months
  * Unstable angina pectoris
  * Hepatocirrhosis
  * Interstitial pneumonia, pulmonary fibrosis, or severe emphysema

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or radiotherapy for colon cancer
* No concurrent radiotherapy
* No concurrent biological response modifiers

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1535 (Actual)
Dates: Start 2008-04; Primary Completion 2012-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Disease-free survival

SECONDARY OUTCOMES:
Overall survival
Adverse event
Pharmaco-economics
Identification of predictive markers

CONTACTS AND LOCATIONS:
Overall Officials: Kenichi Sugihara, MD, PhD, Principal Investigator — Tokyo Medical and Dental University
Locations (1):
- Tokyo Medical and Dental University, Tokyo, Tokyo, Japan

REFERENCES:
- [Derived] Kusumoto T, Ishiguro M, Nakatani E, Yoshida M, Inoue T, Nakamoto Y, Shiomi A, Takagane A, Sunami E, Shinozaki H, Takii Y, Maeda A, Ojima H, Hashida H, Mukaiya M, Yokoyama T, Nakamura M, Munemoto Y, Sugihara K. Updated 5-year survival and exploratory T x N subset analyses of ACTS-CC trial: a randomised controlled trial of S-1 versus tegafur-uracil/leucovorin as adjuvant chemotherapy for stage III colon cancer. ESMO Open. 2018 Oct 7;3(6):e000428. doi: 10.1136/esmoopen-2018-000428. eCollection 2018. PMID 30425843
- [Derived] Yoshida M, Ishiguro M, Ikejiri K, Mochizuki I, Nakamoto Y, Kinugasa Y, Takagane A, Endo T, Shinozaki H, Takii Y, Mochizuki H, Kotake K, Kameoka S, Takahashi K, Watanabe T, Watanabe M, Boku N, Tomita N, Nakatani E, Sugihara K; ACTS-CC study group. S-1 as adjuvant chemotherapy for stage III colon cancer: a randomized phase III study (ACTS-CC trial). Ann Oncol. 2014 Sep;25(9):1743-1749. doi: 10.1093/annonc/mdu232. Epub 2014 Jun 18. PMID 24942277